CLINICAL TRIAL: NCT03760341
Title: Does the Technique of Adenoidectomy Influence the Results of the Surgery? A Prospective Randomized Single Blind Study
Brief Title: Cold Versus Hot Adenoidectomy for Obstructive Sleep Apnea in Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Arie Gordin, MD, Head of pediatric otolaryngology division, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0087-14-RMB
Record Dates: First submitted 2018-11-29; First posted 2018-11-30 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Obstructive Sleep Apnea; Adenoid; Growth
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cold adenoidectomy group (Active Comparator): this group of patient will undergo adenoidectomy by the cold method intervention: adenoidectomy - cold method
  Interventions: Procedure: adenoidectomy - cold method
- hot method adenoidectomy (Active Comparator): this group of patient will undergo adenoidectomy by the cold method intervention: adenoidectomy - hot method
  Interventions: Procedure: adenoidectomy - hot method

INTERVENTIONS:
Procedure: adenoidectomy - cold method — a surgery for adenoid removal or reduction under general anesthesia using surgical curretes
  Arms: cold adenoidectomy group
Procedure: adenoidectomy - hot method — a surgery for adenoid removal or reduction under general anesthesia using suction diathermy
  Arms: hot method adenoidectomy

SUMMARY:
Background: Adenoidectomy is one of the most common procedures done by the otolaryngologist. The procedure can be performed using the cold method (mainly adenoid curettes) or the hot method (suction diathermy). Both techniques have similar intra and post-operative outcomes. However, the long term clinical outcome in improving the sleep disorder symptoms was never compared between the two methods.

Objective: To compare the advantages using the hot method compared to the cold method adenoidectomy in the long term follow up.

Methods: A prospective, randomized, single blinded study of children undergoing adenoidectomy between the years 2014-2017. Patients were randomized to hot or cold adenoidectomy techniques. The primary outcome was change of the Pediatric Sleep Questionnaire Score (PSQ) scores one month and one year after surgery.

DETAILED DESCRIPTION:
The most common cause of sleep disordered breathing in children is enlargement of the adenoids and tonsils relative to the upper airway space.

Obstructive sleep apnea could cause pulmonary and cardiovascular complications, and could influence negatively the l quality of life of the child. Adenoidectomy with or without tonsillectomy is one of the most common procedures done by the otolaryngologist. Adenoidectomy is performed under general anesthesia .The main indications for the procedure include adenoid hypertrophy, obstructive sleep apnea, chronic adenoiditis, and chronic otitis media (ref 1).

Historically recommended instrumentation for performing adenoidectomy has varied from a steel nail, cutting or biting forceps, adenotomes and adenoid curettes.

In 2009 the National institute for health and clinical excellence has published guidelines on the use of suction diathermia adenoidectomy which showed that the method is as effective as or even more than cold method, the method is considered more secure with some advantage in terms of complications of adenoidectomy2, Several studies compared different surgical methods for adenoidectomy. Usually the parameters for comparison were : surgery time, amount of bleeding, complications and regrowth rate (ref 2). None of them examined long term clinical outcome.

The GOLD STANDARD in terms of evaluation of sleep apnea in children is PSG (Polysomnography). However, due to the availability and cost of this test, new methods for assessing these children are studied. Alternatively, some questionnaires were prepared in order to evaluate obstructive sleep apnea in children. One of these questionnaires is the PEDIATRIC SLEEP QUESTIONNARE that contains 22 easy to understand questions which should be answered by YES/NO/IDONT KNOW (ref 3). A result of >0.33 (more than 7 questions answered by yes) should be taken to PSG . In the year 2000 the same group that created the questionnaire published an article in the Sleep Medicine Journal that showed high sensitivity and high validity for sleep apnea diagnosis. The conclusion was that this questionnaire can replace the PSG in clinical trials (ref 3). In 2007 the same group released another study which demonstrates the advantage of the questionnaire compared to PSG evaluation in terms of cognitive and behavioral morbidity of in OSA (Obstructive Sleep Apnea) (ref 4).

In this study the investigators aim to investigate whether there any advantages using SUCTION DIATHERMY in adenoidectomy versus Cold method adenoidectomy in terms of sleep questionnaire score.

ELIGIBILITY:
Inclusion Criteria:

1. age 1 to 15
2. Children with obstructive sleep apnea
3. Children whose parents agreed to be enrolled in the research

Exclusion Criteria:

1. Children who underwent adenoidectomy in the past
2. Refusal for participation by the parent.
3. a diagnosis of malignancy
4. Unable to adhere follow up

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2019-03-20 (Actual)

PRIMARY OUTCOMES:
Pediatric Sleep Questionnaire scores | a month and a year following the surgery
  changes in the Pediatric Sleep Questionnaire scores compared to baseline (before the surgery)

SECONDARY OUTCOMES:
intra-operative complications | intraoperative
  complications during the surgery (i.e. bleeding)
post-operative complications | up till a month following the surgery
  complications following the surgery (i.e. fever, bleeding)

IPD SHARING:
Plan to Share IPD: No